CLINICAL TRIAL: NCT05669365
Title: The Care Ecosystem Consortium Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ochsner Health System (Other); Providence Health & Services (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); HealthPartners Institute (Other); University of Colorado, Denver (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01AG074710 (NIH); 1R01AG074710 (NIH)
Record Dates: First submitted 2022-12-19; First posted 2022-12-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Dementia Alzheimers; Frontotemporal Dementia
MeSH Terms: conditions — Dementia; Dementia, Vascular; Lewy Body Disease; Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care Ecosystem (Experimental): Patient and caregiver dyads receive the Care Ecosystem intervention
  Interventions: Behavioral: Care Ecosystem

INTERVENTIONS:
Behavioral: Care Ecosystem — Applying the principles of person-and-family centered and collaborative care to dementia, the Care Ecosystem (CE) offers proactive, protocol-guided phone- and web-based caregiver support, guidance, and care coordination that extends the reach of dementia primary and specialty care. Care is delivered primarily via the phone and web by unlicensed Care Team Navigators (CTNs), who are trained and supervised by a team of dementia specialists with nursing, social work, and pharmacy expertise. Care Protocols guide proactive, quality care that is documented in the electronic health record (EHR).
  The CTN is an unlicensed, trained dementia care guide who served as the PWD's and caregiver's primary point of contact to the program under nurse supervision. Care team navigators respond to caregivers' immediate needs first, then screen for common problems and provide personalized support and standardized education using the care plan protocols.

SUMMARY:
The Care Ecosystem is an accessible, remotely delivered team-based dementia care model, designed to add value for patients, providers and payers in complex organizational and reimbursement structures. Care is delivered via the phone and web by unlicensed Care Team Navigators, who are trained and supervised by a team of dementia specialists with nursing, social work, and pharmacy expertise. The evidence base to date suggests that the Care Ecosystem improves outcomes important to people with dementia, caregivers, and payers when delivered in a controlled research environment, including reduced emergency department visits, higher quality of life for patients, lower caregiver depression, and reduced potentially inappropriate medication use (Possin et al., 2019; Liu et al., 2022). The investigators propose a rapid pragmatic trial in 6 health systems currently offering the Care Ecosystem program in geographically and culturally diverse populations. The investigators will leverage technology, delivering care via the phone and web and using electronic health records to monitor quality improvements and evaluate outcomes while maximizing external validity. The investigators will evaluate the effectiveness of the Care Ecosystem on outcomes important to patients, caregivers, healthcare providers, and health systems during the pandemic. By evaluating the real-world effectiveness in diverse health systems that are already providing this model of care, this project will bridge the science-practice gap in dementia care during an unprecedented time of heightened strain on family caregivers, healthcare providers and health systems.

DETAILED DESCRIPTION:
This study is a rapid, pragmatic, single-arm trial of 1,275 patients with dementia (PWD) and their caregivers (Total N = 2,550) at 6 US health systems currently offering the Care Ecosystem (CE) intervention to geographically and culturally diverse populations. The investigators will compare the effectiveness of 12-months of the CE intervention with a matched comparison group (N=1,275) identified from the EHR at each site. Patient health care utilization outcomes will be collected via patient insurance / Medicare claims and electronic health record data. Caregiver surveys completed via interview (phone, video or in-person) at baseline, 6-months and 12-months will serve the dual purpose of providing outcome data and supporting care.

This clinical trial is made up of four sub-studies on care quality, utilization, medications, and caregiver and patient experience. While all the sub-studies concern the same intervention group of dyads, each will use data from different sources, different analytic methods, and different controls. Care quality, utilization, and medication metrics will be compared to matched controls identified from the EHR. Caregiver and patient experience metrics will be compared pre/post and to controls from a prior Randomized Control Trial (RCT) (ClinicalTrials.gov NCT02213458). For these reasons, there are primary and secondary endpoints for each.

ELIGIBILITY:
Inclusion criteria, PWD participant

1. Age 18+
2. Provision of verbal consent (or surrogate consent), documented in REDCap, and assent
3. Willingness to enroll in the Care Ecosystem program
4. Lives in the community (i.e., not in an assisted living, board & care, skilled nursing or memory care facility) at the time of enrollment
5. Have a dementia diagnosis documented in the EHR
6. Has had a visit with the referring provider in the last 12 months
7. Has a caregiver with a primary level of responsibility for the patient who is eligible and willing to participate

Inclusion Criteria, Caregiver participant

1. Age 18+
2. Provision of verbal consent, documented in REDCap
3. Has a primary level of responsibility for the care of a PWD-participant who is enrolling in the study
4. Willingness to enroll in the Care Ecosystem program and complete surveys

Exclusion Criteria, PWD participant

1. PWD-participants for whom a substantial amount of the patient's healthcare utilization records cannot be accessed for research purposes by the study team. (see Note)
2. Is currently, or was ever enrolled, in the Care Ecosystem program.
3. Medical documentation indicates that the patient's dementia is a non-progressive type (e.g., due to a head injury or stroke, and not expected to progress).

Note: This exclusion criteria will be operationalized differently at each site based on variations in data access options for their patient population; these options will include EHR and Medicare. A small percentage of participants may be enrolled from underrepresented populations for whom a substantial amount of utilization records cannot be accessed with written approval from the study PI. All participants must be affiliated with one of the 6 participating health systems:

Ochsner Health System Providence Health & Services Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center HealthPartners Institute University of Colorado, Denver University of California, San Francisco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1227 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Dementia Management Quality Measurement Set | Baseline to 12 months
  The rate of completion of a 10-item, adapted Dementia Management Quality Measurement Set. This count variable has a range of 0 (no dementia quality care elements completed) to 10 (all dementia quality care elements completed).
Change in emergency department (ED) visits | Baseline to 12 months
  Number of PWD ED visits, using claims and EHRs.
Change in potentially inappropriate medications for dementia or cognitive impairment | Baseline to 12 months
  Number of high-risk medications used, operationalized using the 2019 Beers criteria, using medication lists from the EHR.
Change in caregiver depression | Baseline to 12 months
  Caregiver depression will be measured by the 9-item Patient Health Questionnaire (PHQ-9), ranging from 0-27 points, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change in PWD hospitalizations | Baseline to 12 months
  Number of PWD hospitalizations, using claims and EHRs.
Change in PWD annual bed days | Baseline to 12 months
  Number of PWD inpatient bed days, using claims and EHRs.
Change in central nervous system (CNS) acting medications | Baseline to 12 months
  Number of CNS acting medications to be avoided in persons with dementia, delirium, or a history of falls or fractures according to the 2019 Beers criteria, using medication lists from the EHR.
Change in caregiver burden | Baseline to 12 months
  The Dementia Burden Scale-Caregiver (DBS-CG) is a composite of the Neuropsychiatric Inventory (NPI-Q) for Distress, the Modified Caregiver Strain Index (MCSI), and and 8-item Patient Health Questionnaire (PHQ-8) with items transformed linearly to be on a 0-100 possible range and then averaged with higher scores indicating higher caregiver burden (Peipert et al., 2018).
Change in caregiver self-efficacy | Baseline to 12 months
  Caregiver self-efficacy score, as measured by a four-item survey with scores ranging from 5-20 points and higher scores indicating higher self-efficacy (Possin et al., 2019; Merrilees et al., 2018).
Change in caregiver anxiety | Baseline to 12 months
  Caregiver anxiety score, as measured by the Generalized Anxiety Disorder 2-item questionnaire (GAD-2), with scores ranging from 0-6 and higher scores indicating higher anxiety.

OTHER OUTCOMES:
Modifications of anti-dementia medications | Baseline to 12 months
  Binary indicator of whether or not a participant's use of anti-dementia medications changed (i.e., started, stopped, or changed treatment with an acetylcholinesterase inhibitor, donepezil, galantamine, rivastigmine, and/or N-methyl-D-aspartate (NMDA) receptor antagonist, memantine).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Possin, PhD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - LA County Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health, Denver, Colorado
  - Ochsner Medical Center, New Orleans, Louisiana
  - HealthPartners, Saint Paul, Minnesota
  - Providence Health, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Investigators will submit resource requests for archived data through a Qualtrics-based form, which will include a signed "Data Use Agreement". These will be reviewed monthly by the investigators. If a request is approved, the study staff will review the requested dataset to ensure it is de-identified and encrypted for transfer, along with a data dictionary.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests will be accepted starting 12 months after study close with no end date.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: http://memory.ucsf.edu/care-ecosystem

REFERENCES:
- [Background] Peipert JD, Jennings LA, Hays RD, Wenger NS, Keeler E, Reuben DB. A Composite Measure of Caregiver Burden in Dementia: The Dementia Burden Scale-Caregiver. J Am Geriatr Soc. 2018 Sep;66(9):1785-1789. doi: 10.1111/jgs.15502. Epub 2018 Aug 10. PMID 30094817
- [Background] Possin KL, Merrilees JJ, Dulaney S, Bonasera SJ, Chiong W, Lee K, Hooper SM, Allen IE, Braley T, Bernstein A, Rosa TD, Harrison K, Begert-Hellings H, Kornak J, Kahn JG, Naasan G, Lanata S, Clark AM, Chodos A, Gearhart R, Ritchie C, Miller BL. Effect of Collaborative Dementia Care via Telephone and Internet on Quality of Life, Caregiver Well-being, and Health Care Use: The Care Ecosystem Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1658-1667. doi: 10.1001/jamainternmed.2019.4101. PMID 31566651
- [Background] Merrilees JJ, Bernstein A, Dulaney S, Heunis J, Walker R, Rah E, Choi J, Gawlas K, Carroll S, Ong P, Feuer J, Braley T, Clark AM, Lee K, Chiong W, Bonasera SJ, Miller BL, Possin KL. The Care Ecosystem: Promoting self-efficacy among dementia family caregivers. Dementia (London). 2020 Aug;19(6):1955-1973. doi: 10.1177/1471301218814121. Epub 2018 Nov 29. PMID 30497302
- [Background] Liu AK, Possin KL, Cook KM, Lynch S, Dulaney S, Merrilees JJ, Braley T, Kiekhofer RE, Bonasera SJ, Allen IE, Chiong W, Clark AM, Feuer J, Ewalt J, Guterman EL, Gearhart R, Miller BL, Lee KP. Effect of collaborative dementia care on potentially inappropriate medication use: Outcomes from the Care Ecosystem randomized clinical trial. Alzheimers Dement. 2023 May;19(5):1865-1875. doi: 10.1002/alz.12808. Epub 2022 Nov 4. PMID 36331050